CLINICAL TRIAL: NCT03331419
Title: Sex Differences in Exercise-related Post-exertional Malaise in ME/CFS
Brief Title: Exercise-related Post-exertional Malaise
Acronym: CFS/ME
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Stony Brook University (Other)
Responsible Party: Sponsor
Other Study IDs: 3R01NR015850-02S1 (NIH)
Record Dates: First submitted 2017-09-22; First posted 2017-11-06 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Chronic Fatigue Syndrome
MeSH Terms: conditions — Fatigue Syndrome, Chronic | interventions — Exercise Test

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Males with Chronic Fatigue Syndrome: Two brief high effort exercise tests on consecutive days in our laboratory in order to provoke abnormalities in ME/CFS patients with respect to autonomic function, symptom exacerbation, and activity limitations.
  Interventions: Behavioral: Exercise test
- Females with Chronic Fatigue Syndrome: Two brief high effort exercise tests on consecutive days in our laboratory in order to provoke abnormalities in ME/CFS patients with respect to autonomic function, symptom exacerbation, and activity limitations.
  Interventions: Behavioral: Exercise test

INTERVENTIONS:
Behavioral: Exercise test — 30 sec of knee squats followed by a six minute walk test repeated on consecutive days.

SUMMARY:
This pilot study is intended to identify sex differences in myalgic encephalomyelitis/ chronic fatigue syndrome (ME/CFS) during recovery from brief but high effort exercise tests. It is expected that women with ME/CFS as compared to males with ME/CFS will show slower recovery from exercise with respect to heart rate and blood pressure, physical functioning, and symptom severity. Also females with ME/CFS as compared to males with ME/CFS will show greater negative impacts on heart rate, blood pressure, physical functioning and symptom severity after the two exercise tests. The findings will have implications for sex differences in the pathophysiology of post-exertional malaise and activity/exercise self-management recommendations, given the expected detrimental effects of the brief intense exercise tests on patients with ME/CFS.

DETAILED DESCRIPTION:
This supplement to the parent study, Myalgic Encephalomyelitis/ Chronic Fatigue Syndrome (ME/CFS): Activity patterns and autonomic function, is intended to enhance the larger home-based study with a face-to-face laboratory arm. Specifically, the investigators propose a pilot study to assess biobehavioral sex differences in ME/CFS during recovery after a brief high exertion exercise task, i.e., a six-minute walk test repeated on two consecutive days. The investigators expect adverse symptomatic, functional, and autonomic effects following this repeat exercise test. This "post-exertional malaise (PEM)" and its impact on global outcomes is a unique feature of ME/CFS that is being studied in the parent observational study conducted by participants entirely in their homes. In the proposed supplement, PEM and its impacts will be captured in real time under controlled conditions in the research team's laboratory. Of particular interest, autonomic effects of PEM on heart function and blood pressure using non-invasive research grade monitors. The specific aims are as follows:

Specific Aim 1: After two high-effort six minute walk tests conducted on consecutive days, female subjects with ME/CFS as compared to male ME/CFS subjects will show slower recovery with respect to cardiovascular autonomic functioning, physical functioning, and symptom resolution. Specific Aim 2: Female subjects with ME/CFS as compared to males with ME/CFS will show greater adverse impact on autonomic and physical functioning and symptom severity after the day 2 exercise test.

To more accurately characterize exercise recovery abnormalities differentiated by sex, the investigators propose to longitudinally monitor symptoms, activity levels, and autonomic status during the week before (baseline) as compared to the week after (follow-up) the two exercise tests. This pilot study will also provide potential cross-validation of the parent project which hypothesizes specific relationships between autonomic function symptom severity and activity limitations. A parallel analysis of sex differences will also be carried out on the data collected in the parent project.

The pilot study will remain within the scope of the original aims of the parent study to identify biobehavioral factors related to PEM, symptom-worsening activity patterns, and non-improvement in ME/CFS. This supplement will expand the parent project's home-based data collection to a controlled setting with direct observation and verification of exercise tests carried out by participants in the principal investigator's laboratory.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 18-65 of both sexes who are considered physically capable of doing and blood pressure monitors (10 min/day) and an actigraph (16 days; waking hours only).
* subjects must meet validated phone-screen eligibility for CFS which will also require the symptom of post-exertional malaise. Also 3 out of 7 secondary symptoms of ME/CFS are required i.e., headaches, tender lymph nodes, sore throat, myalgias, arthralgias, sleep disturbance, and/or problems with memory or concentration.

Exclusion Criteria:

* Cases of fatigue clearly attributable to self-report medical conditions such as untreated hypothyroidism, unstable diabetes mellitus, organ failure, chronic infections, and chronic inflammatory diseases, or AIDS.
* psychiatric disorders include any psychosis, or alcohol/ substance abuse within two years prior to illness onset and any time afterward, and current or past depression with melancholic or psychotic features within 5 years prior to onset of ME/CFS or anytime afterward.
* patients on heart medication or patients not dose-stabilized for at least 3 months on antidepressant drugs
* patients at significant risk of suicide or in need of urgent psychiatric treatment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study sample will be drawn from the population of patients with CFS who (a) respond to local recruitment ads placed online in University announcements and local newspapers; and (b) CFS subjects who have completed the parent study. Ads will emphasize that the study will help to advance our understanding of the biology of CFS (e.g., autonomic functioning).
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2017-11 (Estimated); Primary Completion 2018-10 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Heart rate variability | 15 days
  The time and frequency variation in heart rate recorded on a portable heart monitor

SECONDARY OUTCOMES:
Six minute walk distance (m) | 24 hours
  Distance walked on the six minute walk test
Blood pressure | 24 hours
  Blood pressure taken before and after six minute walk tests
Physical activity | 15 days
  The daily physical activity levels measured with an accelerometer
Online web diary | 15 days
  Symptom intensities recorded on online web diary

CONTACTS AND LOCATIONS:
Overall Officials: Fred Friedberg, PhD, Principal Investigator — Stony Brook University
Locations (1):
- Stony Brook University, Stony Brook, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Friedberg F, Adamowicz JL, Bruckenthal P, Milazzo M, Ramjan S, Zhang X, Yang J. Sex differences in post-exercise fatigue and function in myalgic encephalomyelitis/chronic fatigue syndrome. Sci Rep. 2023 Apr 3;13(1):5442. doi: 10.1038/s41598-023-32581-w. PMID 37012343

DOCUMENTS (3):
  • Study Protocol (2017-09-21): https://cdn.clinicaltrials.gov/large-docs/19/NCT03331419/Prot_000.pdf
  • Informed Consent Form (2017-10-04): https://cdn.clinicaltrials.gov/large-docs/19/NCT03331419/ICF_001.pdf
  • Statistical Analysis Plan (2017-10-10): https://cdn.clinicaltrials.gov/large-docs/19/NCT03331419/SAP_002.pdf